CLINICAL TRIAL: NCT01057394
Title: Post-Market Randomized Controlled Trial: Endoscopically- Guided Ablation vs. Radiofrequency Ablation GuideD by Electroanatomical Mapping to Achieve Permanent Pulmonary Vein Isolation (En-GARDE)
Brief Title: Post-Market Randomized Trial: Endoscopically- Guided Ablation vs. Radiofrequency Ablation
Acronym: En-GARDE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor stopped study for business reasons; not for clinical or clinical outcomes reasons.
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-2758
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency Ablation (Active Comparator): PVI using RF ablation
  Interventions: Device: RF PVI Ablation
- Visually Guided Ablation (Experimental): PVI using visually guided ablation with an endoscopic ablation system
  Interventions: Device: Endoscopically guided PVI Ablation

INTERVENTIONS:
Device: Endoscopically guided PVI Ablation — Endoscopically Guided Ablation using the EAS-AC
  Arms: Visually Guided Ablation
Device: RF PVI Ablation — Radiofrequency ablation
  Arms: Radiofrequency Ablation

SUMMARY:
To compare the safety and chronic Pulmonary Vein isolation of 2 ablation types.

1. visually guided ablation (VGA) using the EAS-AC and
2. radiofrequency ablation

DETAILED DESCRIPTION:
The goal of the study was to compare two interventions, visually-guided endoscopic ablation to standard-of-care radiofrequency (RF) ablation. The study was terminated early by the Sponsor for business reasons before any participants were randomized or treated with RF ablation.

ELIGIBILITY:
* Symptomatic, Paroxysmal Atrial Fibrillation (AF)
* 18 to 75 Years of age
* Generally good overall health as determined by multiple criteria
* Willing to participate in a study
* Others

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — The Mount Sinai Hospital, New York City
Locations (2):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Catholic University of the Sacred Heart, Rome, Italy

REFERENCES:
- See also: Related Info — http://www.cardiofocus.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Sponsor stopped the study for business reasons before any participants were enrolled in the RF arm.
Groups:
- Radiofrequency Ablation; Visually Guided Ablation: Endoscopically Guided Ablation: Visually Guided Ablation using the EAS-AC Radiofrequency Ablation
Period: Overall Study
Arm/Group | Radiofrequency Ablation | Visually Guided Ablation
Started | 0 | 21 (21 enrolled participants)
Completed | 0 | 19 (19 treated participants)
Not Completed | 0 | 2
Not completed — Not eligible | 0 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Visually Guided Ablation
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  Czech Republic | 16
  Italy | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate of Permanent Pulmonary Vein Isolation of EAS-AC Compared to EAM Guided Radiofrequency Ablation
Description: Number of initially isolated pulmonary veins that remain isolated at a 3 month remapping. The unit of measure is treated pulmonary veins (PVs).
Time Frame: 3 Months
Population: Of the 21 enrolled participants, 19 were treated participants and 17 of the 19 came back for the 3 month PV remapping and were thus evaluable for effectiveness. This resulted in 46/59 (78%) pulmonary veins being assessed for chronic isolation.
Measure: Number; unit: isolated pulmonary veins
Arm/Group | Number of Chronically Isolated Pulmonary Veins
Number analyzed (Participants) | 17
isolated pulmonary veins | 46

ADVERSE EVENTS:
Time Frame: Up to 3 months after treatment
Arm/Group | Visually Guided Ablation
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visually Guided Ablation (N=19)
Pericardial effusion (Cardiac disorders) | 1 (1)
Groin bleed (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No